CLINICAL TRIAL: NCT00775853
Title: Biomarkers of Risk of Parkinson Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090010; 09-N-0010
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease; Autonomic Nervous System Diseases; Pure Autonomic Failure
Keywords: Biomarkers; Catecholamines; 18F-Fluoro-L-dopa; Fluorodopamine; Parkinson's Disease; Natural History; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease; Autonomic Nervous System Diseases; Pure Autonomic Failure | interventions — 6-fluorodopamine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals at risk for developing PD: Individuals who may be at risk for developing PD because of genetic risk, olfactory dysfunction, symptomatic rapid eye movement sleep behavior disorder, or orthostatic hypotension
  Interventions: Drug: 6-[18F]Fluorodopamine; Drug: 6-[18F]Fluorodopa; Drug: 13N-Ammonia

INTERVENTIONS:
Drug: 6-[18F]Fluorodopamine
Drug: 6-[18F]Fluorodopa
Drug: 13N-Ammonia

SUMMARY:
This study (https://pdrisk.ninds.nih.gov) will determine if people who have risk factors for Parkinson disease (PD) have biomarkers (objective ways to measure a disease process) that show that the disease process is actually going on, and if people who have abnormal biomarkers go on to develop PD during several years of follow-up. Biomarkers of Parkinson disease (PD) might identify people who are healthy now but may develop the disease later in life.

Healthy volunteers and people who have certain risk factors for developing PD who are between 18 and 70 years of age may be eligible for this study. People with the following risk factors are included:

* Family history of PD
* Loss of sense of smell
* Fall in blood pressure when standing up
* REM behavior disorder (a type of sleep disturbance)

Participants undergo the following tests and procedures:

* Screening examination
* Medical and neurological history and physical examination
* Tests or rating scales for movement, sense of smell, mood, attention, fatigue, pain, and thinking.
* Measurement of blood pressure and pulse rate while lying down and then standing up
* Blood draw for genetic testing
* Inpatient testing at the NIH Clinical Center for 2-3 days, including:
* Measurements while blowing against a resistance
* Measurements of blood pressure and pulse rate
* Blood draws for levels of various chemicals
* PET and MRI scanning
* Lumbar puncture (spinal tap)
* Electrocardiogram
* Skin electrical conduction test (test of sweat production)
* Skin and core temperature measurements
* Transcranial ultrasound (sound-wave test of the head)
* Follow-up testing (up to five visits in 18-month intervals) to repeat some of the tests listed above, excluding the genetic testing and spinal tap

DETAILED DESCRIPTION:
Objective: By the time an individual develops motor symptoms or signs of Parkinson disease (PD) the degeneration of nigrostriatal dopaminergic neurons that produces the movement disorder is already advanced. It is important to identify individuals in whom the pathogenetic process is in a preclinical or prodromal phase. Such individuals would be the best candidates for disease modification clinical trials. PD is characterized by the loss of neurons that use catecholamines as the neurotransmitters, both in the brain and heart. This study is designed to test whether, among people with multiple PD risk factors (at least 3 of the following: family history of PD or genetic risk, olfactory dysfunction, dream enactment behavior, orthostatic hypotension), those with biomarkers of central or myocardial catecholaminergic neurodegeneration are diagnosed with motor symptoms and signs of PD within 7.5 years of follow-up, whereas those with the same risk factors but without biomarkers of catecholaminergic neurodegeneration in either the brain or heart are not diagnosed with motor symptoms and signs of PD during follow-up. Results so far from this study have shown that low cerebrospinal fluid (CSF) levels of 3,4-dihydroxyphenylacetic acid (DOPAC, the main neuronal metabolite of the catecholamine dopamine) and of 3,4-dihydroxyphenylanine (DOPA, the precursor of the catecholamines), low myocardial concentrations of 18F-dopamine-derived radioactivity (an index of deficiency of the catecholamine norepinephrine), and low putamen/occipital cortex ratios of 18F-DOPA-derived radioactivity (an index of putamen dopamine deficiency) distinguish at-risk participants who are diagnosed with motor symptoms and signs of PD within 3 years of follow-up. The study is being continued to follow participants with initial biomarkers data who have not yet been diagnosed with PD. In the follow-up phase we plan on answering the following questions: (1) What proportion of at-risk subjects with negative biomarkers at the time of initial testing develop symptoms of PD during 7.5 years of follow-up? (2) What proportion of at-risk subjects with 1 or 2 positive biomarkers at the time of initial testing develop the motor symptoms and signs of PD during 7.5 years of follow-up? (3) In at-risk subjects who convert from negative to positive biomarkers during follow-up, what proportion develop the motor symptoms and signs of PD during the remaining period until 7.5 years of follow-up?

Study Population: The subjects are individuals who may be at risk for developing PD, because of (a) genetic risk i.e., a family history of PD or genotypic abnormalities known to be associated statistically with PD; (b) olfactory dysfunction i.e., decreased ability to distinguish among odors; (c) symptomatic rapid eye movement (REM) sleep behavior disorder (RBD); or (d) orthostatic hypotension. A total of 200 at-risk subjects undergo catecholaminergic biomarker testing by 18F-DOPA brain and 18F-dopamine cardiac scanning. At-risk subjects with positive biomarkers are compared to at-risk subjects without positive biomarkers, in terms of development of PD during follow-up. Up to 20 control subjects are included, to add to a database of normal values for catecholaminergic biomarkers. As of May 2015, accrual was completed, and participants who already have been characterized in terms of risk factors and biomarkers are in the follow-up phase of the study.

Design: The study includes four phases recruitment, screening, laboratory biomarkers testing, and follow-up. Recruitment is by advertisement and a web site questionnaire of self-reported risk. A screening examination is done at the NIH Clinical Center, to confirm risk status. Based on the screening examination results, subjects undergo inpatient clinical laboratory testing, to identify central and peripheral catecholaminergic denervation. Since May 2015, the study has been in the follow-up phase, during which subjects are being re-tested as inpatients approximately every 18 months for a total of up to 5 re-evaluations (90 months, or 7.5 years), to detect the onset of the characteristic movement disorder in PD and follow the status of putamen and myocardial catecholaminergic innervation.

Outcome Measures:

The primary outcome measure is a clinical diagnosis of PD by a Board-certified neurologist who is blinded to risk factor status and the results of catecholaminergic biomarkers testing; or else completing 7.5 years of follow-up without a diagnosis of PD. If PD diagnosed, time to diagnosis. Secondary outcome measures are the results of UPDRS; F-DOPA brain scanning, F-dopamine cardiac scanning; CSF and plasma neurochemicals; neuropsychological rating scales; autonomic function testing, retrospective CSF proteomics; retrospective DNA analyses.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals who report at least 3 of the following 4 risk factors at the protocol-specific website may be invited to the Screening Examination. All subjects must have ability to provide their own consent for participation in the study. Otherwise eligible candidate participants who are taking medications that would interfere with the scientific results may be included, if (1) the medications are held temporarily or safely substituted for, and (2) the medications are held while the participants are inpatients. The prescribing physician will be contacted, with the participant's permission, if withholding or substituting medication is considered.

1. Genetic Risk: A positive family history (one immediate or more than one non-immediate family member with PD) or positive genetic testing (e.g., LRRK2, alpha-synuclein, glucocerebrosidase) satisfies this risk factor criterion.
2. Olfactory Dysfunction: Olfactory dysfunction reported at the protocol-specific website satisfies this criterion. This may be confirmed by the UPSIT sent by mail prior to the Screening Examination.
3. REM Behavior Disorder (RBD): To satisfy this risk factor criterion, the individual must have movements of the body or limbs associated with dreaming and at least one of the following: potentially harmful sleep behavior, dreams that appear to be acted out, and sleep behavior that disrupts sleep continuity.
4. Orthostatic Hypotension (OH): To satisfy this risk factor criterion, the individual reports symptoms of orthostatic hypotension or having orthostatic hypotension at the protocol-specific website. This may be confirmed by orthostatic vital signs prior to the Screening Examination.

EXCLUSION CRITERIA:

1. Age: People younger than 18 years old or older than 70 years old are excluded.
2. Risk: A candidate subject is excluded if, in the judgment of the Principal Investigator, Protocol participation would place the subject at substantially increased acute medical risk. This includes the risks associated with air travel to the NIH. A candidate subject may be excluded from the study if, in the opinion of the Principal Investigator or Clinical Director, the medical risk outweighs the potential scientific benefit. An example of such risk is inability to travel safely to the NIH Clinical Center, in Bethesda, Maryland, due to a neurological disorder associated with frequent falls.
3. Disqualifying Conditions: A candidate subject is excluded if there is a disqualifying condition. Examples of disqualifying conditions are insulin-dependent diabetes, hepatic or renal failure, symptomatic congestive heart failure, severe anemia, psychosis, ventricular arrhythmias, and symptomatic coronary heart disease.

   * Unable to Provide Consent: Persons who are unable to provide their own consent (e.g., due to dementia) are excluded.
   * MRI: Persons who are unable to undergo MRI safely, due to implanted metal, are excluded from the MRI procedure.
   * Safe Travel: A candidate participant is excluded if the person is unable to travel safely to the NIH Clinical Center, in Bethesda, Maryland, such as due to a neurological disorder associated with frequent falls.
4. Medications: A candidate subject is excluded if clinical considerations require continued treatment with a drug likely to interfere with the scientific results. Chronic, ongoing use of drugs such as tricyclic antidepressants that affect the clinical laboratory results exclude candidate subjects. People with known or suspected allergy or hypersensitivity to any test drug are excluded. Candidate subjects are not to discontinue any medications before discussion with the Principal Investigator, Research Nurse, Nurse Practitioner, or Clinical Fellow. Temporary discontinuation of serotonin and norepinephrine reuptake inhibitors (SNRIs) such as venlafaxine (Effexor), duloxetine (Cymbalta), or des-venlafaxine (Pristiq) can result in rapid rebound of depression or anxiety, and so treatment with SNRIs is exclusionary.
5. Herbal Medicines and Dietary Supplements: If a subject wishes to continue herbal medicines or dietary supplements while on study, but a search of the available medical identifies drug effects that are known or expected to interfere with the experimental results, then the subject may be excluded, at the discretion of Principal Investigator
6. Practical Limitations: People in whom we feel it would be difficult to insert a catheter into a vein may be excluded. People who are not expected clinically to tolerate lying still supine during the testing will be excluded.
7. Pregnancy: Pregnant or lactating women are excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects are individuals who may be at risk for developing PD, because of (a) genetic risk i.e., a family history of PD or genotypic abnormalities known to be associated statistically with PD; (b) olfactory dysfunction i.e., decreased ability to distinguish among odors; (c) symptomatic rapid eye movement (REM) sleep behavior disorder (RBD); or (d) orthostatic hypotension.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2009-05-27 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Parkinson Disease Diagnosed | annually within 7.5 years
  The primary objective of this study is to determine whether among people at increased statistical risk for developing PD those with clinical laboratory biomarkers of central or cardiac catecholamine deficiency are diagnosed with PD during follow-up, whereas those without evidence of central or peripheral catecholamine deficiency are not diagnosed with PD during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: David S Goldstein, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldstein DS, Holmes C, Sullivan P, Lopez G, Gelsomino J, Moore S, Isonaka R, Wu T, Sharabi Y. Cardiac noradrenergic deficiency revealed by 18F-dopamine positron emission tomography identifies preclinical central Lewy body diseases. J Clin Invest. 2024 Jan 2;134(1):e172460. doi: 10.1172/JCI172460. PMID 37883190
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-N-0010.html